CLINICAL TRIAL: NCT07258654
Title: Study of Urinary Impact of Spinal Dysraphism in the Pediatric Population
Acronym: SPINA
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC25_0272
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Dysraphism; Open Dysraphism; Closed Dysraphism
Keywords: dysraphism; spina

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dyspraphism
  Interventions: Other: description of the impact

INTERVENTIONS:
Other: description of the impact — Study of urinary and fecal impact of closed and dysraphism in the pediatric population

SUMMARY:
Spinal dysraphisms are defined as a congenital malformation characterized by a defect in the closure of the neural tube in the caudal region. They are divided into two groups: open dysraphisms, where the skin covering is absent; and closed dysraphisms, where the skin abnormality is less obvious and diagnosis is sometimes more difficult. Both open and closed dysraphisms can cause a variety of neurological disorders, including urinary and fecal dysfunction, which is often more severe in open dysraphisms than in closed dysraphisms, which sometimes go unnoticed and may only become symptomatic during growth. As a result, urinary and fecal repercussions in closed dysraphisms are sometimes overlooked, and the literature on this subject remains scarce. The hypothesis is that a better understanding of the urinary and fecal repercussions of closed dysraphisms would allow for more appropriate and standardized follow-up of these children. The main objective of the study is to describe the urinary impact on children with spinal dysraphism, as well as how they are managed.

ELIGIBILITY:
Inclusion Criteria:

* treated or cared for at Angers University Hospital for spinal dysraphism between January 1, 2014, and December 31, 2024

Exclusion Criteria:

* Differential diagnosis of dysraphism

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients will be selected based on their MRI reports specifying a diagnosis of dysraphism or via diagnostic codes and surgical procedures specific to dysraphism.
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of bladder dysfunction | up to 5 years
  rate of bladder dysfunction in children with open or closed dysraphism

SECONDARY OUTCOMES:
Urinary symptoms | up to 5 years
  urinary symptoms described by patients
Fecal symptoms | up to 5 years
  fecal symptoms that may be described by patients
Urinary treatments implemented | up to 5 years
  urinary treatments that may be implemented during follow-up
Fecal treatments implemented | up to 5 years
  fecal treatments that may be implemented during follow-up
Prenatal diagnosis | Baseline
  presence or absence of a prenatal diagnosis
Clinical signs | Baseline
  linical signs that led to the diagnosis of dysraphism
general symptoms | Baseline
  general symptoms that led to the diagnosis of dysraphism

CONTACTS AND LOCATIONS:
Overall Officials: Louise RENOULT, Study Chair — University Hospital, Angers

IPD SHARING:
Plan to Share IPD: Undecided